CLINICAL TRIAL: NCT03820089
Title: Evaluation of TP US Assesment of Women With Prolapse
Brief Title: Evaluation of TP US in Women With Prolapse
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Other Study IDs: prolapse
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Prolapse
MeSH Terms: conditions — Prolapse | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonography TP — TP us will be made to the included women

SUMMARY:
Many women suffers from uterine and vaginal prolapse Usually they suffer from these symotoms in menopause

DETAILED DESCRIPTION:
The most common cause of pelvic organ prolapse is multiple pregnancy and multiparity

ELIGIBILITY:
Inclusion Criteria:

* Women with history of normal delivery Age between 25 to 75 years

Exclusion Criteria:

* women with cesarean deliveries

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females who have pelvic organ prolapse
Study Population: Women who complains from genital prolapse with previous normal deliveries
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
The number of women who will be properly diagnosed with prolapse by TP us | within 2 months
  The accuracy of TP US in diagnosing the prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt